CLINICAL TRIAL: NCT02822872
Title: Relation Between Emotional Stress and Infertility
Acronym: SFT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, Eyal.levy, Obstetric and gynecology resident, Bnai Zion Medical Center
Other Study IDs: 0107-15-BNZ
Record Dates: First submitted 2016-06-28; First posted 2016-07-04 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
Keywords: infertility; stress; scalp hair; cortisol
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Scalp hair
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- infertile couples: couples addressing IVF treatment due to known infertility will fill questionnaire in order to assess their stress level (as mentioned above), after filling the questionnaire scalp hair sample will be taken to assess chronic cortisol secretion.
  during the IVF treatment the stress level will be assessed every 3 month by using the same system (in order to find match between the stress level and cortisol secretion with the fertility treatment

SUMMARY:
Infertile couples who come for evaluation and treatment in IVF unit could be under psychological stress. Many authors in the past suggested that stress itself is one of the factors that directly influence fecundability rate. In couples treated in IVF unit, the investigators aim to measure chronic stress by measuring hair cortisol level (as a marker for chronic cortisol release) and by filling different questionnaires.

DETAILED DESCRIPTION:
Many speculations regarding the decline in human fecundity are believed to be related to environmental factors, including life style. Among many other factors, perceived psychological stress has been suggested to alter both male and female fertility.

There are many ways to asses stress, one of which is done by filling questionnaires. DASS-21, a 21-item questionnaire, is a set of three self-report scales (Depression, anxiety, stress scale). The negative emotional states of depression, anxiety and stress can be measured using DASS21.

Each of the three DASS scales contains 7 items. Each item is rated on a four-point scale of severity. By using DASS scale, stress and anxiety level of the subject can be monitored in different situations in life.

Another way to asses stress can be done by measuring peptides that are secreted in acute and chronic stress, one of them is cortisol.

Cortisol is a glucocorticoid class steroid hormone; it is produced in humans by the zona fasciculate of the adrenal cortex within the adrenal gland. It is quantified as a marker for hypothalamic pituitary adrenal axis reactivity. In humans, cortisol levels are increased in stress, depression, and selected systemic diseases such as Cushing's syndrome as well as in response to low blood-glucose concentration as well as a response to psychosocial stress.

The experience of chronic adversity or stress is well-known to be associated with a range of negative effects on health. A crucial neuroendocrine axis involved in mediating these effects is the hypothalamus pituitary adrenal axis leading to the secretion of the glucocorticoid cortisol.

Measurement of long-term endogenous production of cortisol can be done by taking urine, saliva or serum samples, while each of these measurements has advantages and limitations. All these methods require multiple samples to provide an assessment of cortisol levels over prolonged periods of time and it is important to note that those measures reflect acutely circulating cortisol level or integrated cortisol secretion over the examined sampling period. Another aspect is that acute cortisol level fluctuates markedly depending on many factors such as circadian rhythmicity, acute stress, cigarettes smoking, alcohol, or exercising.

Another strategy is to measure cortisol is a repeated sampling at different time of the day over several days. But, in order for this strategy to be effective, large number of sampling points during the day are needed.

Taking together, real assessment of long term cortisol secretion can be difficult, thus a new technique has been developed using hair. Positive association between hair cortisol and accumulated salivary free cortisol was seen, and it was concluded that hair cortisol reflects long term cortisol secretion.

In infertile couples who come for evaluation facing stressful time that can cause an even more reduction in fecundity, the investigators will measure long term cortisol secretion and understand the effect of stress and cortisol on infertile couples.

ELIGIBILITY:
Inclusion Criteria:

* infertile couples who addressing IVF treatment in the investigators institute.

Exclusion Criteria:

* couple who don't want to precipitate.
* when there isn't hair to sample.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy couple with known infertility from any reason (both male and female pathology and for unknown infertility) who addressing IVF treatment in Bnai zion medical center.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
concentration of scalp hair cortisol level during IVF treatment (nmol/L) | 3 months
  Hair scalp cortisol will be assessed at couples admission to the investigators IVF unit and at 3 months intervals until pregnancy is achieved

SECONDARY OUTCOMES:
stress assessment during IVF treatment by using questionnaire | 3 months
  Stress assessment using questionnaire will be filled by the couples with each of the scalp hair collection (at admission and in 3 months interval until pregnancy is achieved)

CONTACTS AND LOCATIONS:
Overall Officials: Eyal levy, MD, Principal Investigator — Bnai Zion Medical Center

IPD SHARING:
Plan to Share IPD: No